CLINICAL TRIAL: NCT06173245
Title: The Change of Subfoveal Choroidal Thickness After Intravitreal Injection of Ranibizumab and Its Correlation With Visual Acuity in Diabetic Retinopathy
Brief Title: Subfoveal Choroidal Thickness and Visual Acuity After Intravitreal Injection of Ranibizumab in Diabetic Retinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Egyptian Biomedical Research Network (Network)
Responsible Party: Principal Investigator, Ekram Ragab Abdallah, Specialist of Ophthalmology at El-Mabra hospital, Faculty of Medicine, Al-Azhar University, Assiut, Egypt., Egyptian Biomedical Research Network
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MD/AZ.AST./OPH026/2/199/9/2021
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Subfoveal Choroidal Thickness; Intravitreal; Ranibizumab; Visual Acuity; Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intravitreal injection of ranibizumab (Experimental): These patients were received three intravitreal injection of ranibizumab with one month interval.
  Interventions: Procedure: Intravitreal injection of ranibizumab

INTERVENTIONS:
Procedure: Intravitreal injection of ranibizumab — These patients were received three intravitreal injection of ranibizumab with one month interval. 3D-OCT by enhanced depth spectral-domain imaging (EDI-OCT) was done preoperative and a month after every injection.
  All patients recieved topical anesthesia as 0.5 mg/0.05 ml , ranibizumab is injected 4 mm (3.5 mm in Pseudophakia) from the limbus intravitreally (in the lower temporal quadrant) by a needle (27gauge).

SUMMARY:
The aim of this study is to compare subfoveal choroidal thickness (SFCT) and the visual status before and after intravitreal injection of ranibizumab in diabetic macular edema (DME) with the use of 3D-OCT by enhanced depth spectral-domain imaging (EDI-OCT) with fixating other factors.

DETAILED DESCRIPTION:
Diabetes is a metabolic disorder affecting the ocular vasculature. Although the principal posterior segment changes in diabetes usually occur in the retinal vasculature, additional changes are also observed in the choroid which provides an important blood supply to the outer retina. Diabetic choroidopathy involves choroidal abnormalities occurring in diabetic patients and may participate in mechanisms that lead to the decrease of visual acuity.

Several studies demonstrated the possibility of imaging of the choroid using spectral-domain OCT. Many studies investigated variation in the choroidal thickness (CT) occurring with changes in age and axial length, or in different ocular diseases, Diabetic macular edema (DME) is a major cause of visual loss in diabetic patients.

OCT (Optical coherence tomography) is a non-invasive imaging technique, that was used to obtain a high definition segments of retina. Lately, EDI (enhanced depth imaging) spectral-domain OCT has been explained. (EDI) program routinely captures a cross sectional picture with the choroid near the zero delay line to enhance sensitivity on the external edge of the choroid.

Functional imaging findings also presented a decrease in choroidal flow of the blood in eyes with diabetic retinopathy.

The current purpose of (EDI-OCT), which employing the enhanced depth of field from the inverted picture by locating the OCT device near to the eye, has helped the researchers to study the anatomic variations in the choroid in diabetic eyes.

ELIGIBILITY:
Inclusion Criteria:

* Age from 50 to 70 years.
* Both sexes.
* Patients suffering from diabetic macular edema (DME).

Exclusion Criteria:

* High myopia more than 6 diopters.
* previous injections or retinal surgery.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Change of subfoveal choroidal thickness (SFCT) | 3 months
  All patients will be scheduled for subfoveal choroidal thickness (SFCT) evaluation on the first month, two month and three months by Optical coherence tomography (OCT).

SECONDARY OUTCOMES:
Change of visual acuity (VA) | 3 months
  Regular measurements of visual acuity (VA) over the evaluation visiting

CONTACTS AND LOCATIONS:
Overall Officials: Ekram R Abd-Allah, Master, Principal Investigator — Ophthalmology Department, Faculty of Medicine-Al-Azhar University - Assiut
Locations (1):
- Al-Azhar University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.